CLINICAL TRIAL: NCT01437163
Title: The Growth of Human Scalp Hair Mediated By Visible Red Light Laser and LED Sources.
Brief Title: Treatment of Androgenetic Alopecia in Males and Females
Acronym: LLLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apira Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ApiraTH655
Record Dates: First submitted 2011-09-18; First posted 2011-09-20 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Red Incandescent light source (Sham Comparator)
  Interventions: Device: Laser and/or Light Hair Rejuvenation System
- TopHat 655 (Active Comparator)
  Interventions: Device: TopHat 655 rejuvenation system

INTERVENTIONS:
Device: TopHat 655 rejuvenation system — TopHat 655 system is to be applied every other day for 16 weeks for a pre-programmed time period
  Arms: TopHat 655
Device: Laser and/or Light Hair Rejuvenation System — A red incandescent light source replaces all lasers and light emitting diodes.
  Arms: Red Incandescent light source

SUMMARY:
The purpose of this study is to evaluate the efficacy of Low Level Laser and Light Therapy system configured in a novel product called the TopHat 655 system, for promoting hair growth in males and females diagnosed with androgenetic alopecia of the head.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of androgenetic alopecia
* Fitzpatrick Skin Phototypes I-IV
* Norwood-Hamilton IIa to V for males and Ludwig I or II for females
* Active hair loss within the last 12 months
* Willingness to refrain from using all other hair growth products or treatments
* In overall general good health as determined by the physician investigator

Exclusion Criteria:

* Photosensitivity to laser light and non-laser LED light operating at 655nms.
* Malignancy in the target treatment area
* Other forms of alopecia of the head
* Past medical history of a collagen-vascular disease, thyroid disease or other cutaneous or systemic disease that seriously effects the scalp
* Unwillingness to remove hair replacement products during the therapy sessions
* Using any medications deemed to inhibit hair growth as determined by the physician investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Percentage Increase of Terminal Hairs from Pre-treatment, Baseline Count | After 16 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Raymond J. Lanzafame, MD, Study Director — Raymond J. Lanzafame, MD; Peter S. Halperin, MD, Principal Investigator — Peter S. Halperin, MD; Adolfo Fernandez-Obregon, MD, Principal Investigator — Adolfo Fernandez-Obregon, MD; Jeffrey A Sklar, MD, Principal Investigator — Center for Aesthetic Dermatology
Locations (4):
- United States (4):
  - Adolfo Fernandez-Obregon, MD, Hoboken, New Jersey
  - Peter S. Halperin, MD, New York, New York
  - Raymond J. Lanzafame, MD, Rochester, New York
  - Jeffrey A. Sklar, MD, Woodbury, New York

REFERENCES:
- [Derived] Lanzafame RJ, Blanche RR, Chiacchierini RP, Kazmirek ER, Sklar JA. The growth of human scalp hair in females using visible red light laser and LED sources. Lasers Surg Med. 2014 Oct;46(8):601-7. doi: 10.1002/lsm.22277. Epub 2014 Aug 13. PMID 25124964
- [Derived] Lanzafame RJ, Blanche RR, Bodian AB, Chiacchierini RP, Fernandez-Obregon A, Kazmirek ER. The growth of human scalp hair mediated by visible red light laser and LED sources in males. Lasers Surg Med. 2013 Oct;45(8):487-95. doi: 10.1002/lsm.22173. PMID 24078483